CLINICAL TRIAL: NCT02115087
Title: The Effect of Ultrasound Guided Rectus Sheath Block on Postoperative Analgesia After Laparotomy With Transverse Incision in Children
Brief Title: Efficacy Study of Rectus Sheath Block to Control Postoperative Pain
Acronym: UGRSB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ersel GULEC, Assist.Prof., Cukurova University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UGRSB-123
Record Dates: First submitted 2014-04-09; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Pain, Postoperative
Keywords: laparotomy; levobupivacaine; patient controlled analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound guided rectus sheath block (Experimental): Ultrasound guided rectus sheath block
  Interventions: Procedure: ultrasound guided rectus sheath block
- iv morphine (Active Comparator): 0.1 mg.kg-1 loading dose of morphine by intravenous route in intraoperative period
  Interventions: Drug: Morphine

INTERVENTIONS:
Procedure: ultrasound guided rectus sheath block — the application of rectus sheath block with ultrasound guidance
  Other Names: US guided rectus sheath block
  Arms: ultrasound guided rectus sheath block
Drug: Morphine
  Arms: iv morphine

SUMMARY:
The aim of this study is to evaluate the effect of the ultrasound guided rectus sheath block (RSB) on both intraoperative sevoflurane consumption and postoperative analgesia.

DETAILED DESCRIPTION:
Prospective, randomized study.Forty patients with American Society of Anaesthesiologists (ASA) I-II physical status, aged 3-15 years.Patients are randomly allocated into two groups and are administered general anesthesia and before the beginning of surgery ultrasound guided RSB with 0.2 ml.kg-1, 0.25% of levobupivacaine and thirty minutes before the surgery the loading dose of morphine of 0.1 mg.kg-1 intravenously are received in group RSB and group M, respectively. Patient controlled analgesia (PCA) device with 0.01 mg.kg-1 bolus dose of morphine and 30 minutes lockout interval is set up postoperatively in both groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* 3-15 years of age children
* Abdominal surgery including liver, gall bladder, spleen, small intestine, cecum, colon, rectum, intra-abdominal masses, umbilical, paraumbilical, and inguinal hernia with transverse incision

Exclusion Criteria:

* ASA physical status III and above
* Parents who did not consider to participate in the study
* Having systemic (septicemia, bacteremia) or local infection, bleeding and shock, predisposition for bleeding and anticoagulant therapy given, central nervous system disease, allergy to local anesthetics, severe respiratory, hepatic, and renal failure

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the FLACC scale | Twenty-four hours
  FLACC scale has been used to measure postoperative pain level in children

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ozcengiz, Prof., Principal Investigator — Department of Anesthesiology, Cukurova University Faculty of Medicine
Locations (1):
- Department of Anesthesiology, Cukurova University Faculty of Medicine, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Gelfand HJ, Ouanes JP, Lesley MR, Ko PS, Murphy JD, Sumida SM, Isaac GR, Kumar K, Wu CL. Analgesic efficacy of ultrasound-guided regional anesthesia: a meta-analysis. J Clin Anesth. 2011 Mar;23(2):90-6. doi: 10.1016/j.jclinane.2010.12.005. PMID 21377070